CLINICAL TRIAL: NCT05127278
Title: E-Detection Tool for Emerging Mental Disorders
Acronym: ENTER
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: 885; 215793/Z/19/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Psychosis
Keywords: Ultra High Risk for Psychosis; Clinical High Rish for Psychosis; At Risk Mental State
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Psychosis is a severe mental disorder that involves abnormal experiences and altered behaviour. Although the onset of psychosis occurs in young people, most cases will only be identified later in the course of illness. The delayed detection is the main cause of significant negative long-term outcomes.

The current proposal will develop an innovative E-mental health detection tool to effectively improve the identification of young people with emerging psychosis. This tool will be implemented on digital platforms including websites, tablets and mobile phones. Young people will be asked to complete an online questionnaire and two short online-exercises and will then be invited for face-to-face assessments to further confirm whether they are experiencing an emerging psychosis. This digital approach leverages previous expertise by the research team and it is expected to provide novel avenues to enable the identification of young people with emerging psychosis.

DETAILED DESCRIPTION:
The current proposal will develop an innovative E-DetectioN Tool for Emerging Mental DisoRders (ENTER). This tool will be implemented on a website and the Investigators will invite participants to the site via email-invitations, flyers as well as through advertisements on social media as in previous work byt he team. ENTER will be tested in young people who are experiencing potentially an emerging psychosis, specifically who may meet At Risk Mental State (ARMS) or First Episode Psychosis criteria. The proposed digital approach leverages previous expertise by the research team, and it is expected to provide novel avenues to enable the identification of young people with emerging psychosis. This will ultimately improve the mental health and the life of many young people.

The refined digital screening will enhance previous approaches by incorporating novel features beyond the standard PQ-16 questionnaire, which encompass three overarching domains:

Firstly the Investigators will assess robust epidemiologically-based environmental risk and protective factors that are predicting the onset of psychotic disorders. Some of these factors have already demonstrated prognostic utility, as highlighted by previous work in this area. The selection of these factors has been informed by robust evidence-based synthesis. Digital assessment of exposure to these factors is collected through a Polyrisk Prognostic Score (PPS). This self-rated questionnaire has previously shown to be feasible and non-distressing for young people, discriminating ARMS individuals from healthy. Since most of these factors have been shown to accumulate in ARMS participants, the Investigators expect that the addition of these environmental risk and protective factors will increase the prognostic accuracy of the tool.

Secondly, the Investigators will measure the frequent subthreshold features which characterise emerging psychotic disorders in terms of bipolar risk. To do so the Investigators will employ self-assessment tools that have recently been validated for young people such as the self-rated Bipolar Prodrome Symptom Scale for patients (BPPS-FP) - a brief self-report measure used to assess symptoms of the prodrome to bipolar disorder in order to screen and identify people for whom further evaluation is indicated.

Thirdly, the Investigators will build on recent evidence indicating that cognitive deficits and speech analysis can be used to better identify emerging psychosis. Impaired performance processing speed is one of the most robust indicators of cognitive impairment in psychosis and predicts transition to psychosis in ARMS populations. The Investigators therefore plan to use the self-rated digit symbol task (DST) to assess speed of processing. Moreover, subtle language abnormalities, such as in semantic features and syntactic complexity, can predict outcomes in ARMS populations. To test this the Investigators plan to acquire speech samples in response to Thematic Apperception Test (TAT) to assess speech anomalies.

ENTER will represent a new integrated, comprehensive, scalable, first-in-class e-detection tool that can be implemented in the community. This is particularly important as only 5% of FEP cases are detected through conventional detection strategies that mostly focus on mental health services. Following the validation of ENTER, the Investigators plan that the resulting tool will be implemented on phones and tablets to allow for testing of emerging psychosis in clinical and non-clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* 12-35 years of age
* Informed consent
* Absence of previous psychotic disorders

Exclusion Criteria:

* <12 or >35 years of age
* An existing psychotic disorder

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: General Popualtion
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Validation of online Screener | 2 years
  Validate self report online screener for psychosis by verification with gold standard

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Glasgow University, Glasgow
  - King's College London, London

IPD SHARING:
Plan to Share IPD: No